CLINICAL TRIAL: NCT02297009
Title: Comparison of the Methylation Pattern of DNA in Buccal Swabs From Different Time Points
Status: Terminated | Type: Observational
Why Stopped: Inactive
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S57170
Record Dates: First submitted 2014-10-31; First posted 2014-11-21 (Estimated); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: DNA Methylation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Buccal cells

GROUPS / COHORTS (1):
- Volunteers: 30 volunteers, half men and half women Buccal swab
  Interventions: Procedure: Buccal swab

INTERVENTIONS:
Procedure: Buccal swab — Buccal swabs will be taken from the volunteers

SUMMARY:
A buccal swab will be taken using a cotton stick by rubbing it against the buccal mucosa. Samples will be taken from the same participant at different timepoints.

DNA will be extracted from the buccal cells on the swabs using a commercial extraction kit and will be quantified by a nano-drop spectrophotometer.

We will determine global and gene-specific methylation and hydroxymethylation alterations by UPLC/MS/MS. Hydrolyzed DNA into individual nucleosides will be analyzed for the quantitative measurement of 5-methylCytosine and 5-hydroxymethylCytosine on Triple Quadrupole UPLC/MS/MS platform. Secondly, specific methylation in the CpG islands of tumor suppressor and promoter genes, and genes involved in the oxidative stress pathways will be assessed by PCR-pyrosequencing.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian

Exclusion Criteria:

-

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Students and research staff
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-12; Primary Completion 2024-07 (Actual); Study Completion 2024-07 (Actual)

PRIMARY OUTCOMES:
%Methylation (%) | 5 weeks

SECONDARY OUTCOMES:
%Hydroxymethylation (%) | 5 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- BIOMAT, Leuven, Belgium